CLINICAL TRIAL: NCT07151443
Title: Comparison of Conventional and Retroclavicular Approaches for Ultrasound-guided Infraclavicular Brachial Plexus Block in Obese Patients
Brief Title: Comparison of Conventional and Retroclavicular Approaches for Ultrasound-guided Infraclavicular Brachial Plexus Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, İbrahim Topcu, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-006
Record Dates: First submitted 2025-02-13; First posted 2025-09-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Nerve Block; Pain Management; Forearm Surgery; Hand Surgery; Upper Extremity
Keywords: Infraclavicular Block; Obesity; Upper Extremity; Hand surgery; Forearm surgery
MeSH Terms: conditions — Agnosia; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional approach to infraclavicular block (Active Comparator): After the patients are monitored and placed in the supine position, after appropriate field sterilization, Conventional approach to infraclavicular block will be performed on the patients using 25 ml of local anesthetic solution (20 ml 0.5% bupivacaine + 5 ml 2% lidocaine) under ultrasound guidance.
  Interventions: Procedure: Conventional approach to infraclavicular block
- Retroclavicular approach to the infraclavicular block (Active Comparator): After the patients are monitored and placed in the supine position, after appropriate field sterilization, Retroclavicular approach to the infraclavicular block will be performed on the patients using 25 ml of local anesthetic solution (20 ml 0.5% bupivacaine + 5 ml 2% lidocaine) under ultrasound guidance.
  Interventions: Procedure: Retroclavicular approach to the infraclavicular block

INTERVENTIONS:
Procedure: Conventional approach to infraclavicular block — Conventional approach to infraclavicular block will be performed on the patients using 20 ml of 0.5% bupivacaine 5ml of %2 lidocaine under ultrasound guidance.
  Arms: Conventional approach to infraclavicular block
Procedure: Retroclavicular approach to the infraclavicular block — Retroclavicular approach to the infraclavicular block will be performed on the patients using 20 ml of 0.5% bupivacaine 5ml of %2 lidocaine under ultrasound guidance.
  Arms: Retroclavicular approach to the infraclavicular block

SUMMARY:
Forearm and hand surgeries are among the most frequently performed surgical interventions both in trauma patients and electively.In these procedures, alternative anesthesia methods such as general anesthesia, regional intravenous anesthesia, regional peripheral nerve blocks and local anesthesia are available.

Peripheral nerve blockade can be used for anesthesia and analgesia.This method allows patients to undergo surgery without general anesthesia and increases patient satisfaction by providing effective analgesia in the postoperative period.

The aim of this study was to compare the conventional and retroclavicular approaches to infraclavicular block in patients undergoing forearm and hand surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-80 years of age
* Those with ASA score II-III
* Those with a body mass index (BMI) >30
* Patients who are suitable for forearm and hand surgery under regional anesthesia in the operating room

Exclusion Criteria:

* Patients who cannot perceive and evaluate pain
* Patients who want to have surgery under general anesthesia
* Patients in whom regional anesthesia is contraindicated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Block Performance Time | During regional anesthesia
  Total block performance time (from skin puncture to needle removal) will be recorded

SECONDARY OUTCOMES:
Pain Score | Up to 24 hours
  Pain will be assessed using a visual analog scale from 0 mm (no pain) to 100 mm (worst pain) at rest and when coughing. Pain assessment will be made at 0, 1, 6, 12, 18, and 24 hours after surgery.
Patient Satisfaction | 1 day
  Quality of recovery-15 (QoR-15) score was used as the satisfaction score. The patient-reported Turkish QoR-15 score includes 15 questions that evaluate the patient's postoperative recovery. The QoR-15 score is grouped under two groups, A and B. A high QoR-15 score, a score between 0 (poor) and 10 (excellent) for each item, and a total score of 150 indicate better quality of recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)